

## HAROKOPIO UNIVERSITY

## SCHOOL OF HEALTH SCIENCE AND EDUCATION DEPARTMENT OF NUTRITION AND DIETETICS

## INFORMED CONSENT FORM TO THE INTERVENTIONTAL STUDY WITH TITLE:

"Effect of a dietary intervention that includes daily consumption of a novel biscuit enriched with Greek edible mushrooms, rich in β-glucans, on intestinal health-related parameters of healthy older adults: a randomized controlled trial"

CODE: (completed by the investigator)

| declare my consent to participate in the interventional research study entitled "Effect of a dietary intervention that includes daily consumption of a novel biscuit enriched with Greek edible mushrooms, rich in $\beta$ -glucans, on intestinal health related parameters of healthy older adults: a randomized controlled trial". Associated Professor of Microbiology in Harokopio University, Dr. Adamantini Kyriacou, is the scientific supervisor of the research. The study aims to evaluate whether the daily consumption, for 3 months, of a novel biscuit enriched with mushroom powder containing 3g of $\beta$ -glucans has an effect on the intestinal microbiota of individuals over 60 years old. |
|---|
| This study includes the evaluation of dietary intake and physical activity, measurements of anthropometric characteristics, the completion of questionnaires (frequency or gastrointestinal symptoms, sleep habits, memory and orientation ability), as well as the sampling of biological samples (blood, urine and feces). Any questions I may have about any study process will be fully answered by those in charge of the study. Any personal information about me and the results of the measurements that will be obtained during the study, will remain confidential. I declare that I sign this Informed Consent Form on my own free will. |
| Subject's Acknowledgement |
| Date: |
| (Subject's signature) |